CLINICAL TRIAL: NCT00196131
Title: Changes in Morphine Handling and Response in Patients With Brain Trauma
Brief Title: Problems With Morphine Use in Patients With a Severe Brain Injury
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dalhousie University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Richard Hall, Dalhousie University
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: Dal05-01; CIHRMOP-74451
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2006-09

CONDITIONS: Head Trauma; Subarachnoid Hemorrhage; Close Head Injury
Keywords: morphine; head injury; SAH
MeSH Terms: conditions — Craniocerebral Trauma; Subarachnoid Hemorrhage; Head Injuries, Closed | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0 (No Intervention)
  Interventions: Drug: morphine

INTERVENTIONS:
Drug: morphine — only patients with a head injury currently receiving Morphine continuously or prm can and have an ICP drain can be enrolled into study

SUMMARY:
Hypothesis: During severe brain trauma (injury, surgery) the ensuing inflammatory response in the central nervous system (CNS) results in a decrease in the expression of the transporter protein p-glycoprotein (PGP) in the blood brain barrier. This loss results in the penetration into the brain of certain drugs that are normally excluded by the transporter protein. In this study the working hypothesis is that the agitation observed in patients with CNS trauma treated with morphine is related to the inflammation evoked loss of PGP in the blood brain barrier and the accumulation of the morphine metabolite 3-morphine glucuronide.

DETAILED DESCRIPTION:
It is well established that the metabolism, distribution and elimination of certain drugs is affected by inflammatory processes. This results from the expression of cytochrome and drug transporter proteins that are altered during the generation of host defense mechanisms. This has major implications in inflammation and infection when the capacity of the liver and other organs to handle drugs are severely compromised. From studies in animals individual cytochrome P450 isozymes and p-glycoprotein (PGP) are down regulated at the level of gene transcription with a resulting decrease in the corresponding mRNA, protein and enzyme/transporter activity. The loss in drug metabolism and transport is channeled predominantly through the production of cytokines which ultimately modify specific transcription factors. Other proposed mechanisms that apply to specific cytochrome P450s involve post translational steps including enzyme modification and increased degradation. When inflammatory responses are confined to the brain there is a loss of cytochrome P450 and PGP not only in the brain but also in peripheral tissues. This involves a yet to be identified mode of signaling between the brain and periphery but it does involve the production of cytokines from a peripheral source.

In clinical medicine there are numerous examples of a decreased capacity to handle drugs during infections and disease states that involve an inflammatory component. This often results in altered drug responses and increased toxicities. Inflammation mediated alterations in the metabolism of endogenous compounds can also lead to altered physiology. Recently it has been shown in rodents that inflammatory responses within the brain alter drug disposition in the brain and in peripheral systems. Of particular note to the use of drugs in patients with a brain trauma is a recent study in our laboratory carried out in rodents showing that the transport of some drugs across the blood brain barrier is dramatically changed during a CNS inflammatory response. The reason this occurs is the loss in expression of the drug transporter protein (PGP). This allows drugs which are normally transported out of the brain by PGP to enter and cause CNS toxicity. Such changes in drug handling capacity during inflammation/infection will continue to be one of the many factors that complicate therapeutics.

In humans with a severe CNS trauma (injury, surgery) an inflammatory response commonly occurs within the brain. It has also been our clinical observation that when these patients receive morphine as part of their care the drug is tolerated for a few days but many patients develop agitation that we believe is related to morphine therapy. Our working hypothesis is that a metabolite of morphine which is a CNS irritant (3-morphine glucuronide) can enter the brain in increased amounts because of the inflammation evoked loss in the transporter protein PGP in the blood brain barrier. In normal circumstances morphine is metabolized in the liver to two major metabolites (3-morphine glucuronide and 6-morphine glucuronide). These metabolites are excluded to some extent by a functioning PGP in the blood brain barrier. If the PGP diminishes in the blood brain barrier as a result of CNS inflammation then these morphine metabolites will increase in concentration in the brain. Some support for this idea can be taken from the recent studies showing that the inhibition of PGP by chemical means increases the concentration of the 6-glucuronide of morphine following the administration of morphine to rats. Although the 6-glucuronide is more potent than morphine with similar actions, the 3-glucuronide is a CNS irritant and may cause the agitation observed in these patients. We propose to measure these metabolites on both sides of the blood brain barrier in patients with CNS trauma/inflammation to determine if the agitation correlates with the build up of metabolites. If we can demonstrate that these metabolites increase in the CNS as a result of inflammation this study will have far reaching consequences to many other drugs that are normally excluded from the brain in this manner (eg digoxin, cyclosporine A, HIV protease inhibitors) during their use in any condition that involves an inflammatory component in the CNS.

ELIGIBILITY:
Inclusion Criteria:

* Sustained a head trauma (closed head injury or subarachnoid hemorrhage [SAH])
* Fitted with a intraventricular drainage catheter
* Currently being treated with morphine

Exclusion Criteria:

* Patient is receiving another PGP inhibitor drug other than morphine or midazolam

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-01; Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
see the ratios of cerebrospinal fluid (CSF)/blood increase with time as the inflammation progresses | prospective

SECONDARY OUTCOMES:
ratios of morphine and its metabolites in CSF and blood with the RASS will determine if observed CNS stimulation occurs at a time when the levels of 3-morphine glucuronide is high on the brain side of the blood brain barrier | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Richard I Hall, MD, Principal Investigator — Capital Health- QE II HSC
Locations (1):
- Capital Health -QE II HSC, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Goralski KB, Hartmann G, Piquette-Miller M, Renton KW. Downregulation of mdr1a expression in the brain and liver during CNS inflammation alters the in vivo disposition of digoxin. Br J Pharmacol. 2003 May;139(1):35-48. doi: 10.1038/sj.bjp.0705227. PMID 12746221